CLINICAL TRIAL: NCT01010191
Title: Pilot Randomized Controlled Trial
Brief Title: Harnessing Placebo Effects: Non-Deceptive Use of Placebo in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Ted Kaptchuk, Harvard Medical School
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16986
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; no organic digestive disease
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellulose pill (Experimental): The active intervention is a sugar pill.
  Interventions: Other: Sugar pill
- No treatment (No Intervention): The control arm is wait list control

INTERVENTIONS:
Other: Sugar pill
  Arms: Cellulose pill

SUMMARY:
Irritable bowel syndrome patients will be given either placebo pill or no treatment for a period of 3 weeks.

DETAILED DESCRIPTION:
Seventy patients with irritable bowel syndrome (IBS) will be randomized to either 1) placebo pill or 2) no treatment and followed for 3 weeks. The study will involve three visits: baseline, midpoint and end point. At baseline all patients will physical examination, be evaluated for IBS and be administered standardized IBS questionnaires including: "IBS adequate relief" questionnaire, IBS global symptom improvement scale, IBS quality of life and IBS symptom severity scale. At midpoint and endpoint the same questionnaires will be administered. Patients on no treatment will be offered education on managing IBS at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome.

Exclusion Criteria:

* Any signs of organic bowel disease such as rectal bleeding.
* No other major illnesses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
IBS Global Improvement Scale | 3 weeks

SECONDARY OUTCOMES:
IBS Adequate Relief | 3 weeks
IBS quality of life (QoL) | 3 weeks
IBS Symptom Severity Scale | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kaptchuk TJ, Friedlander E, Kelley JM, Sanchez MN, Kokkotou E, Singer JP, Kowalczykowski M, Miller FG, Kirsch I, Lembo AJ. Placebos without deception: a randomized controlled trial in irritable bowel syndrome. PLoS One. 2010 Dec 22;5(12):e15591. doi: 10.1371/journal.pone.0015591. PMID 21203519